CLINICAL TRIAL: NCT03311932
Title: A Two-part, Single Centre, Open-label, Randomised, Single Dose, Two-period, Crossover, Relative Bioavailability Study of Infacort® Versus Cortef® in Dexamethasone-suppressed Healthy Adult Male and Female Subjects in the Fasted and Fed States.
Brief Title: A Study of Infacort® Versus Cortef® in Healthy Adult Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: Simbec Research (Industry); Brush Clinical Research Ltd. (Industry); Voet Consulting (Industry); Bionical-Emas Pharma Ltd (Unknown); Medical Matters International Ltd (Industry); Nichol Pharma Services Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Infacort 007
Record Dates: First submitted 2017-07-11; First posted 2017-10-17 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cortef® Tablets - fasted (Active Comparator): Single dose of 20mg Cortef® Tablets - fasted arm
  Interventions: Drug: Cortef®
- Infacort® - fasted (Experimental): Single dose of 20mg Infacort® - fasted arm
  Interventions: Drug: Infacort®
- Cortef® Tablets - fed (Active Comparator): Single dose of 20mg Cortef® Tablets - fed arm
  Interventions: Drug: Cortef®
- Infacort® - fed (Experimental): Single dose of 20mg Infacort® - fed arm
  Interventions: Drug: Infacort®

INTERVENTIONS:
Drug: Infacort® — Immediate release multiparticulate formulation (granules) of hydrocortisone
  Arms: Infacort® - fasted; Infacort® - fed
Drug: Cortef® — Immediate release hydrocortisone tablets
  Arms: Cortef® Tablets - fasted; Cortef® Tablets - fed

SUMMARY:
This was a two-part, single centre, open-label, randomised, single dose, two-period, crossover study to evaluate the bioavailability of Infacort® versus Cortef® immediate release hydrocortisone tablets in dexamethasone-suppressed healthy adult male and female subjects in the fasted and fed states.

DETAILED DESCRIPTION:
The study was conducted in two parts (Part 1 and 2) which were not performed sequentially. In Part 1, 26 subjects were dosed in a fasted condition and in Part 2, 25 subjects were dosed in a fed condition. Each part comprised of a pre-study screen, followed by 2 treatment periods (1 and 2) and a post-study follow-up.

Screening assessments (for Parts 1 and 2) were conducted within the 28 days before the first administration of a study intervention. Eligible participants were asked to return for the 2 treatment periods. Continued eligibility was confirmed pre-dose for each treatment period.

Part 1 (fasted state): Treatment Periods: Eligible participants received a single dose of each study intervention over 2 treatment periods (1 per treatment period). Each treatment period was approximately 1.5 days in duration. Participants arrived at the Clinical Unit on Day -1 and dexamethasone 1 mg was administrated at approximately 22:00 hours and then again at approximately 06:00 and 12:00 of Day 0 of each treatment period to suppress endogenous cortisol production. The study intervention was administered at approximately 08:00 on Day 0 in the fasted state (after an overnight fast of at least 10 hours). Participants were discharged following the 12-hour post-dose blood sampling and consumption of a snack (Day 0).

Part 2 (fed state): The same procedures were followed as for Part 1 except that study interventions were administered in a fed condition (30 minutes after the start of a standardised high-fat breakfast). PK samples in both study parts were collected pre-dose and up to 12 hours post-dose (19 samples for each treatment period) for measurement of cortisol levels. Safety was evaluated throughout the study. There was at least a 7-day washout period (up to a maximum of 14 days) between dose administrations. After completion of both study periods, participants were to return 7±2 days later for a final follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females between 18 and 55 years of age, inclusive (at screening).
2. A body mass index (BMI) of 18 to 30 kg/m2 (inclusive)
3. No clinically significant abnormal serum biochemistry, haematology or urine examination values, as defined by the Investigator.
4. A negative urinary drugs of abuse screen. A positive alcohol test or drugs of abuse test could be repeated at the discretion of the Investigator.
5. Negative human immunodeficiency virus (HIV) and hepatitis B and C test results.
6. No clinically significant abnormalities in the 12-lead ECG, as defined by the Investigator.
7. No clinically significant deviation outside of the normal ranges for blood pressure and heart rate measurements, as defined by the Investigator.
8. Male participants (unless anatomically sterile or abstinence from sexual intercourse was in line with preferred and usual lifestyle) and sexual partners were to use an effective contraception method during the study and for 3 months after the last intervention, for example:

   * Established use of oral, injected or implanted hormonal contraceptive.
   * Intrauterine device or intrauterine system.
   * Condom and diaphragm with spermicide.
9. Female participants of childbearing potential (unless abstinence from sexual intercourse was in line with preferred and usual lifestyle) with a negative pregnancy test at screening and on admission, and willing to use an effective method of contraception from the first dose until 3 months after the last intervention, for example:

   * Established use of oral / injected / implanted hormonal methods of contraception.
   * Intrauterine device or intrauterine system.
   * Barrier methods: condom + occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
10. Female participants of non-childbearing potential with negative pregnancy test at screening. For the purposes of the study, non-childbearing was defined as being amenorrhoeic for at least 12 consecutive months or at least 4 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy). Menopausal status was confirmed at screening by demonstrating that levels of follicle stimulating hormone (FSH) fell within the respective reference range. In the event a participant's menopausal status had been clearly established (for example, the participant indicated she had been amenorrhoeic for 10 years) but FSH levels were not consistent with a post-menopausal condition, determination of eligibility was at the Investigator's discretion following consultation with the Sponsor.
11. Participants were available to complete both study periods and the follow-up visit.
12. Participants satisfied a medical examiner that they were fit to participate in the study.
13. Participants were able to read and understand the ICF and provide written informed consent to take part in the study.

Exclusion Criteria:

1. A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
2. Receipt of any medication other than acetaminophen within the 14 days prior to dosing (including topical steroids, vitamins, dietary supplements or herbal remedies).
3. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
4. Receipt of any vaccination within the previous one month.
5. Presence of infections (systemic fungal and viral infections, acute bacterial infections).
6. Current or previous history of tuberculosis.
7. A clinically significant history of previous allergy/sensitivity to hydrocortisone and/or dexamethasone.
8. Meeting any of the contraindications for Cortef® and/or dexamethasone, as detailed in the USPI and Summary of Product Characteristics (SmPC).
9. A clinically significant history of drug or alcohol abuse.
10. Inability to communicate well with the Investigator (i.e. language problem, poor mental development or impaired cerebral function).
11. Participation in a New Chemical Entity or marketed drug clinical study within the previous 3 months or, five half-lives of study drug, whichever is the longer period. (NB. the three-month washout period between trials is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
12. Participants who had consumed more than 2 units of alcohol per day within the 7 days prior to the first dose or had consumed any alcohol within the 48-hour period prior to the first dose.
13. Donation or receipt of equal to or greater than 450 mL of blood within the previous three months.
14. Participants who smoked (or ex-smokers who had smoked within the 6 months prior to the first dose). This included e-cigarette and shisha users.
15. Participants who worked shifts (i.e. regularly alternated between days, afternoons and nights).
16. Vegetarians, vegans or those with other dietary restrictions which meant they were unable to consume the standardised high-fat breakfast (applicable to Part 2 only).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters for serum cortisol - Maximum serum concentration (Cmax) | Blood samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 and 12 hours; in both periods
  Comparing the maximum serum cortisol concentration (Cmax) of Infacort® compared to Cortef® immediate release hydrocortisone tablets.This PK endpoint will be derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
Pharmacokinetic parameters for serum cortisol - Area under the serum cortisol concentration-time curve (AUC0-t) | Blood samples taken at 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5 , 6, 8, 10 and 12 hours; in both periods
  Comparing the total drug exposure over time for Infacort® compared to Cortef®. This PK endpoint will be derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
Pharmacokinetic parameters for serum cortisol - Area under the curve extrapolated to infinity (AUC0-inf) | Blood samples taken at 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5 , 6, 8, 10 and 12 hours; in both periods
  Comparing the total drug exposure over time for Infacort® compared to Cortef® extrapolated to infinity from dosing time, based on the last observed concentration. This This PK endpoint will be derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.

SECONDARY OUTCOMES:
Adverse events (AEs) | Through study completion - approximately 6 weeks
  AEs observed throughout the study
Vital signs | Through study completion - approximately 6 weeks
  Observed changes in vital signs data during the course of the study
Electrocardiogram (ECG) | Through study completion - approximately 6 weeks
  Observed changes in ECG data during the course of the study
Safety Laboratory Data | Through study completion - approximately 6 weeks
  Observed changes in Safety Laboratory data during the course of the study
Pharmacokinetic parameters for serum cortisol - Time to maximum cortisol concentration (Tmax) | Blood samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 and 12 hours; in both periods
  This PK endpoint will be derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
Pharmacokinetic parameters for serum cortisol - Elimination rate constant (Kel) | Blood samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 and 12 hours; in both periods
  This PK endpoint will be derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
Pharmacokinetic parameters for serum cortisol - Terminal half life (t 1/2) | Blood samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 and 12 hours; in both periods
  This PK endpoint will be derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
Pharmacokinetic parameters for serum cortisol - Serum cortisol clearance (CL/F) | Blood samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 and 12 hours; in both periods
  Calculated as Dose / AUC0-inf. This PK endpoint will be derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
Pharmacokinetic parameters for serum cortisol - Distribution during terminal elimination (Vz/F) | Blood samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 and 12 hours; in both periods
  Volume of distribution based on the terminal elimination phase following extravascular administration derived from baseline adjusted and unadjusted serum cortisol.

CONTACTS AND LOCATIONS:
Overall Officials: A Koch, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd., Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No